CLINICAL TRIAL: NCT03148431
Title: A Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of LY3002815 in Healthy Subjects
Brief Title: A Study of LY3002815 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to business decisions
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16529; I9G-MC-CCBA (Other: Eli Lilly and Company); 2016-004453-33 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3002815 (Experimental): Escalating doses of LY3002815 administered intravenously (IV) once in healthy participants
  Interventions: Drug: LY3002815
- Placebo (Placebo Comparator): Placebo administered IV once in healthy participants
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3002815 — Administered IV
  Arms: LY3002815
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The purposes of this study are to determine:

* The safety of the study drug and any side effects that might be associated with it.
* How much of the study drug gets into the blood stream and how long it takes the body to remove it in healthy participants.

Participants will be admitted to the Clinical Research Unit (CRU) for 3 overnight stays.

This study involves a single dose of LY3002815 or placebo given as an injection into the vein. This study will last approximately 16 weeks including screening. Additional follow-up may be required.

This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination. Males will be required to use reliable method of birth control. Females have to be of non-child-bearing potential
* Have a body mass index (BMI) of 18 to 32 kilograms per meter squared (kg/m²) inclusive, at screening

Exclusion Criteria:

* Have family history of early onset Alzheimer's Disease (AD)
* Have impaired cognitive function
* Have significant abnormalities in brain magnetic resonance imaging (MRI); or have contraindications for MRI
* Have significant allergic reactions to LY3002815, or related compounds, or have significant allergies to humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone
* Women who are lactating
* Have clinically significant neurological or psychological illness, or other illnesses that could affect the study results

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through at least 85 days after administration of study drug

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3002815 | Baseline through at least 85 days after administration of study drug
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of LY3002815 | Baseline through at least 85 days after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, UK, United Kingdom